CLINICAL TRIAL: NCT05619133
Title: Effects and Underlying Mechanisms of Photobiomodulation (PBM) on Health and Well-Being
Brief Title: PBM Effects on Health and Well-being in Humans
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Seaborough Life Science B.V. (Industry)
Collaborators: Chrono@Work B.V. (Unknown); University of Groningen (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Basic Science
Other Study IDs: PBM2022
Record Dates: First submitted 2022-11-01; First posted 2022-11-16 (Actual); Last update posted 2022-11-16 (Actual); Status verified 2022-11

CONDITIONS: Sleep Deprivation; Circadian Rhythm Disorders
MeSH Terms: conditions — Sleep Deprivation; Chronobiology Disorders

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (5):
- placebo (No Intervention): No PBM will be emitted from the device; dose: 0 J.cm-2
- PBM High standard (Experimental): A PBM high standard dose of 6.5 J.cm-2 with a wavelength of 850 nm, a pulse of 15 Hz and 8 ms and duty factor of 12%
  Interventions: Device: PBM
- PBM High wavelength (Experimental): A PBM high dose of 6.5 J.cm-2 with a wavelength of 940 nm, a pulse of 15 Hz and 8 ms and duty factor of 12%
  Interventions: Device: PBM
- PBM High pulse (Experimental): A PBM high dose of 6.5 J.cm-2 with a wavelength of 850 nm, a pulse of 100 Hz and 1.2 ms and duty factor of 12%
  Interventions: Device: PBM
- PBM High skin only (Experimental): A PBM high standard dose of 6.5 J.cm-2 with a wavelength of 850 nm, a pulse of 15 Hz and 8 ms and duty factor of 12%, but in this case the participants will wear filtering googles which will not allow PBM from entering the eyes
  Interventions: Device: PBM

INTERVENTIONS:
Device: PBM — In this study, the health benefits of the addition of NIR to the light spectrum of a desk lamp already available in the market will be investigate; Ikea Ypeperlig, to which a module with high power Lumileds NIR-Leds will be attached with beam angle of 90 degrees. They will be attached in such a way that, when the lamp is installed in the right place, a 1sr beam that covers the users face, neck and hands and lower arms on the desk with the required intensity of 5mW/cm2 of NIR at the skin surface.
  The device will be equipped with 3 sensors:
  1. A distance sensor connected to the driver of the NIR-leds, such that when the user leans forward or backward, the intensity of the NIR is automatically adjusted such that the intensity on the skin remains 5mW/cm2 (see figure below).
  2. a presence sensor
  3. ambient vertical lux sensor by which amount of light that enters the users' eye will be measured since it is known that these have an effect sleep, mood and performance.
  Arms: PBM High pulse; PBM High skin only; PBM High standard; PBM High wavelength

SUMMARY:
The goal of this clinical study is to assess the effects of different photobiomodulation (PBM) conditions in men and women between 25 and 65 years old with daytime sleepiness/drowsiness and /or mild mood complaints but be otherwise healthy. The main question it aims to answer are:

1. Does PBM significantly affect health and well-being?
2. Are PBM effects wavelength dependent?
3. Are PBM effects pulse dependent?
4. Are the eyes needed to assert an PBM effect or is exposure only to the skin sufficient?
5. What are the cellular, metabolic pathways underlying the systemic effects of PBM.

Participants will have to:

1. Exposed themselves 5 times per week during 2 weeks to the PBM stimuli between 9:30 and 12:30.
2. A week before the baseline measurement, participants will have to start wearing a Fitbit Versa 3, and will have to continuously wear until the end of the study.
3. In the afternoon of the baseline day as well as in the afternoons after 5 and 10 PBM sessions (week 1 and week 2, respectively), participants will have to go to the lab for blood withdraw.
4. In the evening of the baseline day as well as in the evenings after 5 and 10 PBM sessions (week 1 and week 2, respectively), participants will have to collect saliva samples as well as to complete questionnaires.

It will be a double-blind placebo-controlled field study with a between subject comparison.

DETAILED DESCRIPTION:
Five conditions (groups) will be tested:

Dose (J.cm-2) Wavelength (nm) Pulse (Hz,ms) Duty factor Area Cond 1 6.5 850 15, 8 12% Skin + eyes Cond 2 6.5 940 15, 8 12% Skin + eyes Cond 3 6.5 850 100, 1 12% Skin + eyes Cond 4 0 850 15, 8 12% Skin + eyes Cond 5 6.5 850 15, 8 12% Skin

ELIGIBILITY:
Inclusion Criteria:

Healthy, no chronic disease

* Age between 25 - 65 years.
* Suffer from daytime sleepiness/drowsiness and or a mild mood disturbance (ESS >5 or BDI equal to or higher than 13 but lower than 20, PSQI > 5)
* Participants will have to have a desk type of work and/or have 3 hours per day between 9:30 am and 12:30 at their office/home in which they could sit in front of the lamp.

Exclusion Criteria:

Depressive mood (BDI -II > 20)

* Pregnancy
* Menopause symptoms
* Drug use during the last three months known to interfere with sleep, alertness, the biological clock and/or light sensitivity (i.e. regular usage of sleep medication or stimulating substances)
* Use of immune suppressants. High levels of caffeine intake during a day (5 or more cups, according to https://www.voedingscentrum.nl/encyclopedie/cafeine.aspx#blok7, there are no negative effects expected from 4 caffeine products in normal adults)
* High alcohol intake (more than 4 for men and more than 3 for women, drinks per day) for more than 5 days in the past month, including binge drinking and heavy drinking according to https://www.niaaa.nih.gov/publications/brochures-and- fact-sheets/alcohol-facts-and-statistics.
* Participant is not able to refrain from using recreational drugs during the 4 weeks of the study.
* Shift work schedule in the 3 months prior to participation and/or planned during the 2 weeks of the study
* Environmental factors in everyday life that may disturb sleep and cannot be prohibited (e.g. young children, noisy environment)
* Travel over 2 or more time zones in the month prior to participation
* Travel to sunny holiday locations/wintersports 1 month before participation
* Personal plans that prevent them for using the intervention during 2 consecutive weeks

Ages: 25 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2023-01-01 (Estimated); Primary Completion 2023-05-31 (Estimated); Study Completion 2023-05-31 (Estimated)

PRIMARY OUTCOMES:
Change from baseline in subjective mood after 5 and after 10 PBM sessions | Baseline, after 2 weeks, after 4 weeks
  Mood VAS scale, 0-10, higher score means better
Change from baseline in subjective drowsiness after 5 and after 10 PBM sessions | Baseline, after 2 weeks, after 4 weeks
  Epworth Sleepiness Scale, 0-24, higher score means worse
Change from baseline in depressions scale after 5 and after 10 PBM sessions | Baseline, after 2 weeks, after 4 weeks
  Beck Depression Inventory Second Edition, 0-63, higher score means worse
Change from baseline in general activation after 5 and after 10 PBM sessions | Baseline, after 2 weeks, after 4 weeks
  Activation-Deactivation check list, 5-20, higher score means better
Change from baseline in deactivation after 5 and after 10 PBM sessions | Baseline, after 2 weeks, after 4 weeks
  Activation-Deactivation check list, 11-14, higher score means worse
Change from baseline in high activation after 5 and after 10 PBM sessions | Baseline, after 2 weeks, after 4 weeks
  Activation-Deactivation check list, 5-20, higher score means worse
Change from baseline in general deactivation after 5 and after 10 PBM sessions | Baseline, after 2 weeks, after 4 weeks
  Activation-Deactivation check list, 5-20, higher score means worse
Change from baseline in subjective sleep quality scores after 5 and after 10 PBM sessions | Baseline, after 2 weeks, after 4 weeks
  Pittsburgh Sleep quality scale, 0-21, higher score means worse
Change from baseline in resting heart rate after 5 and after 10 PBM sessions | Through study completion
  Fitbit Versa 3
Change from baseline in objective sleep quality scores after 5 and after 10 PBM sessions | Through study completion
  Fitbit Versa 3
Change from baseline in IFN- gamma concentrations after 5 and after 10 PBM sessions | Baseline, after 2 weeks, after 4 weeks
  Blood
Change from baseline in TNF-alpha concentrations after 5 and after 10 PBM sessions | Baseline, after 2 weeks, after 4 weeks
  Blood
Change from baseline in TGF-beta1concentrations after 5 and after 10 PBM sessions | Baseline, after 2 weeks, after 4 weeks
  Blood
Change from baseline in il-1 concentrations after 5 and after 10 PBM sessions | Baseline, after 2 weeks, after 4 weeks
  Blood
Change from baseline in il-6 concentrations after 5 and after 10 PBM sessions | Baseline, after 2 weeks, after 4 weeks
  Blood
Shift from baseline in dim light melatonin onset after 5 and after 10 PBM sessions | Baseline, after 2 weeks, after 4 weeks
  Saliva
Change from baseline in cortisol levels at bedtime after 5 and after 10 PBM sessions | Baseline, after 2 weeks, after 4 weeks
  Saliva
Change from baseline in targeted metabolomics concentration after 5 and after 10 PBM sessions | Baseline, after 4 weeks
  Blood

CONTACTS AND LOCATIONS:
Overall Officials: Marijke Gordijn, PhD, Principal Investigator — Chrono@Work

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Fulop AM, Dhimmer S, Deluca JR, Johanson DD, Lenz RV, Patel KB, Douris PC, Enwemeka CS. A meta-analysis of the efficacy of laser phototherapy on pain relief. Clin J Pain. 2010 Oct;26(8):729-36. doi: 10.1097/AJP.0b013e3181f09713. PMID 20842007
- [Result] Heiskanen V, Pfiffner M, Partonen T. Sunlight and health: shifting the focus from vitamin D3 to photobiomodulation by red and near-infrared light. Ageing Res Rev. 2020 Aug;61:101089. doi: 10.1016/j.arr.2020.101089. Epub 2020 May 25. PMID 32464190
- [Result] Liebert A, Bicknell B, Markman W, Kiat H. A Potential Role for Photobiomodulation Therapy in Disease Treatment and Prevention in the Era of COVID-19. Aging Dis. 2020 Dec 1;11(6):1352-1362. doi: 10.14336/AD.2020.0901. eCollection 2020 Dec. PMID 33269093
- [Result] Miranda-Silva W, Gomes-Silva W, Zadik Y, Yarom N, Al-Azri AR, Hong CHL, Ariyawardana A, Saunders DP, Correa ME, Arany PR, Bowen J, Cheng KKF, Tissing WJE, Bossi P, Elad S; Mucositis Study Group of the Multinational Association of Supportive Care in Cancer / International Society for Oral Oncology (MASCC/ISOO). MASCC/ISOO clinical practice guidelines for the management of mucositis: sub-analysis of current interventions for the management of oral mucositis in pediatric cancer patients. Support Care Cancer. 2021 Jul;29(7):3539-3562. doi: 10.1007/s00520-020-05803-4. Epub 2020 Nov 6. PMID 33156403